CLINICAL TRIAL: NCT04246307
Title: Investigation of Systemic and Regional Haemostasis During Liver Transplantation by Comparing ClotPro® and TEG ® Viscoelastic Tests
Brief Title: Investigation of Systemic and Regional Haemostasis During Liver Transplantation by Comparing ClotPro® and TEG®
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Semmelweis University (Other)
Collaborators: DiaCare Solution Kft (Unknown)
Responsible Party: Principal Investigator, Janos Fazakas MD, PhD, Associate Professor, Semmelweis University
Other Study IDs: ETT-TUKEB 20325-2/2019
Record Dates: First submitted 2019-12-30; First posted 2020-01-29 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Haemostasis Disorders
Keywords: end-stage liver disease; liver transplantation; bleeding management; coagulopathy; thromboelastography; viscoelastic coagulation monitoring; thromboeleastometry; ClotPro
MeSH Terms: conditions — End Stage Liver Disease; Hemostatic Disorders | interventions — Thrombelastography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: TEG® and ClotPro® parameters — Systemic sampling is performed six times:
  * before the surgery (S1)
  * during the hepatectomy, 10 minutes before the anhepatic phase (S2)
  * in the anhepatic phase, before starting portal vein anastomosis: (S3)
  * in the neohepatic phase, 15 minutes after releasing portal vein clamping: (S4)
  * in the neohepatic phase, at the end of the surgery: (S5)
  Regional sampling from the portal vein representing afferent flow to the liver is performed once:
  • in the anhepatic phase, before starting portal vein anastomosis: (R)
  Simultaneously with haemostasis and blood gas analyses, the following investigations will be performed (the following tests are also routinely performed at the given time points, independently of this study):
  * haemodynamic measurements by PiCCO
  * arterial blood gas analysis from radial artery catheter
  * central venous blood gas analysis from subclavian vein catheter
  * blood temperature measurement in the femoral artery by PiCCO catheter
  * hourly urinary output
  Other Names: Intreventional

SUMMARY:
The purpose of the research is to compare the global and the portal haemostasis during liver transplantation by functional investigations using TEG® and ClotPro® tests. The study aims at revealing important coagulation-associated links affecting the outcome of the liver transplant surgery.

DETAILED DESCRIPTION:
Donor data Liver donor data are investigated following the "Donor Query" used for donor reports of the Organ Coordination Office of the Hungarian National Blood Transfusion Service. (http://www.ovsz.hu/sites/ovsz.hu/files/szervadomanyozas_dokumentum/donacio/donorlekerdezo-2013-06-03.pdf) The donor is identified by the alarm ID and the Eurotransplant number (ETnr). Independently of this study, the "Donor Query" is completed for all donor reports and helps to asses donor suitability.

Recipient preoperative data In case of a liver alarm, age, body metrics, medical history, type and severity of hepatic disease, concomitant diseases, and admission laboratory test results of the recipient are recorded. Independently of this study, these data/procedures are recorded/performed for all liver transplant candidates.

Surgical data In addition to technical data of the surgery, data on intraoperative fluid balance, transfusion need, supportive therapy (vasopressor or inotropic therapy, renal replacement therapy), and number and indication of any reoperation are also recorded.

Intraoperative sampling times and investigations

During a liver transplantation, independently of this study, the following procedures are performed to monitor the patient's haemodynamics, homeostasis, and haemostasis:

* femoral artery catheterisation by pulse index contour cardiac output (PiCCO) catheter - haemodynamic monitoring by PiCCO
* radial artery catheterisation - arterial blood gas and arterial pressure monitoring
* subclavian or internal jugular vein catheterisation - central venous pressure (CVP) and central venous blood gas monitoring, drug administration
* external jugular vein catheterisation - blood sampling for haemostasis tests (TEG® and ClotPro® conventional laboratory tests - international normalized ratio (INR), activated partial thromboplastin time (aPTT), fibrinogen, antithrombin (AT), factor V (FV), factor VII (FVII), factor X (FX), factor XIII (FXIII)
* 2 3 large peripheral veins - fluid resuscitation
* permanent urinary catheter - hourly urine output

During the study, for the analysis of haemostasis (TEG®, ClotPro®) and blood gases, 3.5 ml blood will be sampled per site and time from the external jugular vein catheter representing the systemic sample and from the portal vein representing the regional sample. Before performing the portal vein anastomosis, a small amount of blood is routinely flushed from the portal vein. Regional blood sampling is performed from this blood.

Systemic sampling is performed five times:

* before the surgery (S1)
* during the hepatectomy, 10 minutes before the anhepatic phase (S2)
* in the anhepatic phase, before starting portal vein anastomosis: (S3)
* in the neohepatic phase, 15 minutes after releasing portal vein clamping: (S4)
* in the neohepatic phase, at the end of the surgery: (S5)

Regional sampling from the portal vein is performed once:

• in the anhepatic phase, before starting portal vein anastomosis: (R)

Simultaneously with haemostasis and blood gas analyses, the following investigations will be performed (as the part of the anaesthesia protocol):

* haemodynamic measurements by PiCCO
* arterial blood gas analysis from radial artery catheter
* central venous blood gas analysis from subclavian vein catheter
* blood temperature measurement in the femoral artery by PiCCO catheter
* hourly urinary output Postoperative phase and follow-up In the immediate postoperative phase, postoperative heamodynamic, pulmonary, renal function, liver graft function) and their supportive therapy will be analysed.

Laboratory tests (quantitative and qualitative blood count, INR, aPTT, fibrinogen, AT, FV, FVII, FX, FXIII, C reactive protein (CRP), procalcitonin (PCT), electrolytes, creatinine, urea, bilirubin, liver enzymes, albumin, total protein, immunosuppressive drug levels) will be performed at the end of the surgery, at postoperative hours 12 and 24, on postoperative days 2, 3 and 7. As far as possible these tests will be carried out on day 30 and one year after the surgery as well.

Vasopressor and inotropic therapies will be analysed. The duration of assisted ventilation and the presence of pleural fluid or any sign of postoperative pneumonia will be evaluated. Urinary output as well as need for renal replacement therapy and the modality of that will also be investigated. Liver graft function will be monitored by means of laboratory parameters and graft perfusion with sonography. Initial poor function (IPF) and primary nonfunction (PNF) During the study, one-year graft and patient survival rates, the occurrence of small bile duct complications associated with arterial perfusion disorders, and the recurrence of underlying hepatic disease will be recorded. If a biopsy is taken within one year, histopathological results will also be evaluated.

Methodology and organisation of the study Informing patients on the study will occur during liver alarms by an anaesthesiologist. One copy each of the Patient Information Leaflet and the Informed Consent Form signed by the patient, the consenting physician and the principal investigator will be given to the patient. A copy of each of them will be filed in the medical records of the patient and the original one will be part of the research documentation.

During the study, tests for the investigation of parameters described in the protocol will be performed by the patients' physicians and other health care professionals involved in patient care.

Coagulation tests During the study, viscoelastic tests will be performed by TEG® and ClotPro® instruments.

Blood sampling for systemic TEG® and ClotPro® tests will be performed from the routinely catheterised external jugular vein while blood for regional tests will be taken from the portal vein of the recipient. After obtaining informed consent from the patient, 3.5 mL of blood samples will be collected in citrate tubes designated for the study at surgery phases described above. Investigations will be conducted by a TEG® 5000 thromboelastograph (Haemonetics Corp., Switzerland) and a ClotPro® (enicor GmbH, Germany) analyser. Results will subsequently be analysed by computed statistical tests. Simultaneously with viscoelastic tests, blood gas analyses will also be performed from the collected blood samples to obtain current pH, pCO2, and bicarbonate and calcium levels and their role in coagulation will be considered for the study. Furthermore, central body temperature will also be continuously monitored and recorded during the perioperative phase.

During TEG® and ClotPro® measurements in this study, the following parameters will be compared:

for TEG®, the following parameters will be considered in the study: R (reaction time): fluid phase of coagulation, time to formation of 2 mm clot; K (kinetics): time to formation of 20 mm clot; α: angle between 2 mm and 20 mm clot; MA (maximum amplitude): ultimate size of the clot; Ly30: percent rate of lysis at 30 minutes post MA. During the liver transplantation citrated kaolin test (CK-TEG) will be completed.

for ClotPro®, the following parameters will be considered in the study: CT (clotting time): indicates the fluid phase of coagulation (corresponds to R in TEG®); CFT (clot formation time): coagulation kinetics parameter, time between formation of 2 mm and 20 mm clot (corresponds to K in TEG®); α: angle (slope) of line between CT and CFT; A10 and A20 describe clot size (amplitude) at certain time points; MCF (maximum clot firmness): represents the ultimate size (maximum amplitude) of the clot (corresponds to MA in TEG®); clot lysis index at 30 (CLI30) describes the ratio between the maximum clot firmness and the amplitude 30 minutes after clotting time, LT (lysis time): characterises tPA effect.

During the liver transplantation EX-test, IN-test, FIB-test, TPA-test, RVV-test, and ECA-test tests will be completed.

Blood gas analyses Analyses are currently done by a GEM® PremierTM 3500 instrument. The blood gas analyser measures the following parameters: pH, pCO2, pO2, sodium, potassium, ionised calcium, blood glucose, lactate, bicarbonate, base excess, haemoglobin, haematocrit. Blood gas analyses are performed from the arterial and central vein samples. From the portal vein, blood sample is collected by the surgeon.

Laboratory parameters The following parameters will be measured at the laboratory by Sysmex CS 2000i, Sysmex XN-1000 (Sysmex Europe GmbH, Hungary) and Dimension® RxL Max® Integrated Chemistry System (Siemens Healthcare GmbH, Hungary)

* quantitative and qualitative blood count
* INR, aPTT, fibrinogen, AT, FV, FVII, FX, FXIII, sodium, potassium, magnesium, phosphate, ionised calcium
* creatinine, urea
* CRP, PCT
* total and direct bilirubin
* albumin
* liver enzymes: alkaline phosphatase (ALP), glutamic-oxaloacetic transaminase (GOT), glutamate-pyruvate transaminase (GPT), gamma-glutamyltransferase (GGT), lactate dehydrogenase (LDH), cholinesterase
* pancreatic enzymes: amylase, lipase Time of each laboratory test is determined by the study protocol. Laboratory tests associated with this study do not differ from the current clinical practice and thus, pose no additional interventions over the standard care.

Haemodynamic parameters Haemodynamic monitoring is performed for all patients undergoing liver transplantation in the perioperative period, independently from this study. Monitoring is done by a PiCCO instrument. During thermodilution measurements, cardiac output (CO), cardiac index (CI), intrathoracic blood volume index (ITBI), extravascular lung water index (EVLWI), stroke volume (SV), stroke volume variation (SVV), cardiac function index (CFI), maximum left ventricular contractility (dPmax), and mean arterial pressure (MAP) will be monitored.

CVP will be monitored via the catheterised subclavian vein. Time of each haemodynamic test is determined by the study protocol. Haemodynamic tests associated with this study do not differ from the current clinical practice and thus, pose no additional interventions over the standard care.

Oxygen delivery and consumption Parameters characterising oxygen delivery (oxygen delivery index; DO2I) and consumption (oxygen consumption index; VO2I) are calculated from arterial and central venous blood gas analysis results and from haemodynamic parameters.

Statistical methods Statistical analyses will be performed by Social Sciences software (SPSS; SPSS Inc, Chicago, Illinois, USA).

Continuous and discrete variables will be analysed by independent samples t tests (two categories) and one-way analyses of variance (one-way ANOVA; more categories), respectively. Two continuous variables will be compared by Spearman's rank correlation test. Discrete variables will be tested by Pearson's Chi squared test. Ordinary variables will be compared by Mann-Whitney U test or Kruskal-Wallis test. For multivariate analyses, logistic regression models will be generated.

Significance level will be set to 5% (p ≤ 0.05).

ELIGIBILITY:
Inclusion criteria:

* Patients requiring liver transplantation for chronic liver failure are to be enrolled at time of their liver transplantation.
* Patients ≥18 years of age at the time of liver transplantation.
* Liver transplantation will be performed between January 1st 2020 and January 1st 2021

Exclusion criteria:

* acute liver failure
* Failure to obtain informed consent from the patient.
* Patients <18 years of age.
* Patients lacking legal competence.
* Coagulation tests included in the study protocol cannot be performed for any technical reason or samples cannot be collected.
* Combined liver and kidney transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring liver transplantation for hepatic failure are to be enrolled at time of their liver transplantation.
  Patients ≥18 years of age at the time of liver transplantation.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between TEG® and ClotPro® parameters | 24 hours
  If there is correlation between TEG® and ClotPro® parameters:
  1. reaction time (R) in citrated kaolin TEG (CK-TEG) and clotting time (CT) in IN-test (ClotPro®)
  2. kinetics (K) in CK-TEG and clot formation time (CFT) in IN-test
  3. Alpha-angel in CK-TEG and IN-test
  4. maximum amplitudo (MA) in CK-TEG and maximum clot firmness (MCF) in IN-test
  5. percent rate of lysis (Ly30) in CK-TEG and clot lyzis index (CLI30) in IN-test

SECONDARY OUTCOMES:
Difference between systemic and the portal haemostasis | 24 hours
  If there is a significant difference between the systemic and the portal haemostasis before graft reperfusion:
  1. R, K, Alpha-angel, MA, MCF and Ly30 in CK-TEG from systemic and portal sample
  2. CT, CFT, Alpha-angel, MCF, CLI30 in EX-test, IN-test, FIB-test, TPA-test, RVV-est, ECA-test from systemic and portal sample
  3. Conventional laboratory tests: international normalized ratio (INR), activated partial thromboplastin time (aPTT), fibrinogen, antithrombin (AT), factor V (FV), factor VII (FVII), factor X (FX), factor XIII (FXIII) from systemic and portal sample
  4. Blood gas analysis: pH, pCO2, pO2, sodium, potassium, ionised calcium, blood glucose, lactate, bicarbonate, base excess, haemoglobin, haematocrit from systemic and portal sample
Correlation between the fetures of the intraoperative systemic and regional haemostasis and severity of the liver disease | 24 hours
  1. Child-Turcotte-Pugh (CTP) score and CK-TEG (R, K, Alpha-angel, MA, MCF and Ly30) parameters from systemic and systemic samples
  2. CTP score and ClotPro (CT, CFT, Alpha-angel, MCF, CLI30 in EX-test, IN-test, FIB-test, TPA-test, RVV-est, ECA-test) parameters from systemic and portal samples
  3. Model for End-stage Liver Disease (MELD) score and CK-TEG (R, K, Alpha-angel, MA, MCF and Ly30) parameters from global and systemic samples
  4. MELD score and ClotPro (CT, CFT, Alpha-angel, MCF, CLI30 in EX-test, IN-test, FIB-test, TPA-test, RVV-est, ECA-test) parameters from systemic and portal samples
  5. MELD-Na score and CK-TEG (R, K, Alpha-angel, MA, MCF and Ly30) parameters from systemic and portal samples
  6. MELD-Na score and ClotPro (CT, CFT, Alpha-angel, MCF, CLI30 in EX-test, IN-test, FIB-test, TPA-test, RVV-est, ECA-test) parameters from systemic and portal samples
Correlation between local and systemic haemostasis and any subsequent coagulopathic or thrombotic complications | 24 hours
  If there is a correlation between local and systemic haemostasis and any subsequent coagulopathic or thrombotic complications (reoperation for haemorrhage, portal vein or hepatic artery thrombosis).
  1. Need for reoperation due to haemorrhage and CK-TEG (R, K, Alpha-angel, MA, MCF and Ly30) parameters from systemic and portal samples
  2. Need for reoperation due to haemorrhage and ClotPro (CT, CFT, Alpha-angel, MCF, CLI30 in EX-test, IN-test, FIB-test, TPA-test, RVV-est, ECA-test) parameters from systemic and portal samples
  3. Need for reoperation due to portal vein or hepatic artery thrombosis and CK-TEG (R, K, Alpha-angel, MA, MCF and Ly30) parameters from systemic and portal samples
  4. Need for reoperation due to portal vein or hepatic artery thrombosis and ClotPro (CT, CFT, Alpha-angel, MCF, CLI30 in EX-test, IN-test, FIB-test, TPA-test, RVV-est, ECA-test) parameters from systemic and portal samples

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University, Budapest, Pest County, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adams MJ, Irish AB, Watts GF, Oostryck R, Dogra GK. Hypercoagulability in chronic kidney disease is associated with coagulation activation but not endothelial function. Thromb Res. 2008;123(2):374-80. doi: 10.1016/j.thromres.2008.03.024. Epub 2008 May 16. PMID 18486198
- [Background] Agarwal B, Wright G, Gatt A, Riddell A, Vemala V, Mallett S, Chowdary P, Davenport A, Jalan R, Burroughs A. Evaluation of coagulation abnormalities in acute liver failure. J Hepatol. 2012 Oct;57(4):780-6. doi: 10.1016/j.jhep.2012.06.020. Epub 2012 Jun 23. PMID 22735303
- [Background] Aird WC. Phenotypic heterogeneity of the endothelium: I. Structure, function, and mechanisms. Circ Res. 2007 Feb 2;100(2):158-73. doi: 10.1161/01.RES.0000255691.76142.4a. PMID 17272818
- [Background] Aird WC. Phenotypic heterogeneity of the endothelium: II. Representative vascular beds. Circ Res. 2007 Feb 2;100(2):174-90. doi: 10.1161/01.RES.0000255690.03436.ae. PMID 17272819
- [Background] Aird WC. Spatial and temporal dynamics of the endothelium. J Thromb Haemost. 2005 Jul;3(7):1392-406. doi: 10.1111/j.1538-7836.2005.01328.x. Epub 2005 May 9. PMID 15892866
- [Background] Aird WC. Vascular bed-specific hemostasis: role of endothelium in sepsis pathogenesis. Crit Care Med. 2001 Jul;29(7 Suppl):S28-34; discussion S34-5. doi: 10.1097/00003246-200107001-00013. PMID 11445731
- [Background] Akkina SK, Asrani SK, Peng Y, Stock P, Kim WR, Israni AK. Development of organ-specific donor risk indices. Liver Transpl. 2012 Apr;18(4):395-404. doi: 10.1002/lt.23398. PMID 22287036
- [Background] American Society of Anesthesiologists Task Force on Perioperative Blood Transfusion and Adjuvant Therapies. Practice guidelines for perioperative blood transfusion and adjuvant therapies: an updated report by the American Society of Anesthesiologists Task Force on Perioperative Blood Transfusion and Adjuvant Therapies. Anesthesiology. 2006 Jul;105(1):198-208. doi: 10.1097/00000542-200607000-00030. No abstract available. PMID 16810012
- [Background] Babik B, Blaskó Gy, Fazakas J, et al.: Az életveszélyes perioperatív vérzések ellátása: szakmai irányelv. Aneszteziológia és Intenzív Terápia. 2013, 43(3): 113-143.
- [Background] Bischof D, Dalbert S, Zollinger A, Ganter MT, Hofer CK. Thrombelastography in the surgical patient. Minerva Anestesiol. 2010 Feb;76(2):131-7. Epub 2009 Nov 24. PMID 20150854
- [Background] Bolliger D, Gorlinger K, Tanaka KA. Pathophysiology and treatment of coagulopathy in massive hemorrhage and hemodilution. Anesthesiology. 2010 Nov;113(5):1205-19. doi: 10.1097/ALN.0b013e3181f22b5a. PMID 20881594
- [Background] Scarpelini S, Rhind SG, Nascimento B, Tien H, Shek PN, Peng HT, Huang H, Pinto R, Speers V, Reis M, Rizoli SB. Normal range values for thromboelastography in healthy adult volunteers. Braz J Med Biol Res. 2009 Dec;42(12):1210-7. doi: 10.1590/s0100-879x2009001200015. Epub 2009 Oct 30. PMID 19882085
- [Background] Colomina MJ, Diez Lobo A, Garutti I, Gomez-Luque A, Llau JV, Pita E. Perioperative use of prothrombin complex concentrates. Minerva Anestesiol. 2012 Mar;78(3):358-68. PMID 22357373
- [Background] Dalmau A, Sabate A, Aparicio I. Hemostasis and coagulation monitoring and management during liver transplantation. Curr Opin Organ Transplant. 2009 Jun;14(3):286-90. doi: 10.1097/MOT.0b013e32832a6b7c. PMID 19300254
- [Background] Dirkmann D, Hanke AA, Gorlinger K, Peters J. Hypothermia and acidosis synergistically impair coagulation in human whole blood. Anesth Analg. 2008 Jun;106(6):1627-32. doi: 10.1213/ane.0b013e31817340ad. PMID 18499589
- [Background] Durila M, Malosek M. Rotational thromboelastometry along with thromboelastography plays a critical role in the management of traumatic bleeding. Am J Emerg Med. 2014 Mar;32(3):288.e1-3. doi: 10.1016/j.ajem.2013.09.038. Epub 2013 Oct 2. PMID 24286666
- [Background] Edelberg JM, Christie PD, Rosenberg RD. Regulation of vascular bed-specific prothrombotic potential. Circ Res. 2001 Jul 20;89(2):117-24. doi: 10.1161/hh1401.093954. PMID 11463717
- [Background] Fazakas J, Smudla A: Véralvadás zavarok kritikus állapotú betegekben. In Bogár L, Molnár Zs (szerk.): Az intenzív terápia gyakorlata. Budapest, Medicina, 2013, 432-442.
- [Background] Feng S, Goodrich NP, Bragg-Gresham JL, Dykstra DM, Punch JD, DebRoy MA, Greenstein SM, Merion RM. Characteristics associated with liver graft failure: the concept of a donor risk index. Am J Transplant. 2006 Apr;6(4):783-90. doi: 10.1111/j.1600-6143.2006.01242.x. PMID 16539636
- [Background] Gando S, Wada H, Thachil J; Scientific and Standardization Committee on DIC of the International Society on Thrombosis and Haemostasis (ISTH). Differentiating disseminated intravascular coagulation (DIC) with the fibrinolytic phenotype from coagulopathy of trauma and acute coagulopathy of trauma-shock (COT/ACOTS). J Thromb Haemost. 2013 May;11(5):826-35. doi: 10.1111/jth.12190. PMID 23522358
- [Background] Ganter MT, Spahn DR. Perioperative coagulation management. Best Pract Res Clin Anaesthesiol. 2010 Mar;24(1):vii-viii. doi: 10.1016/j.bpa.2009.10.002. No abstract available. PMID 20402165
- [Background] Girardis M, Marietta M. Hemostasis in acute liver and kidney failure: nothing is as it seems. Kidney Int. 2013 Jul;84(1):22-4. doi: 10.1038/ki.2013.121. PMID 23812363
- [Background] Hunt BJ. Bleeding and coagulopathies in critical care. N Engl J Med. 2014 Feb 27;370(9):847-59. doi: 10.1056/NEJMra1208626. No abstract available. PMID 24571757
- [Background] Innerhofer P, Kienast J. Principles of perioperative coagulopathy. Best Pract Res Clin Anaesthesiol. 2010 Mar;24(1):1-14. doi: 10.1016/j.bpa.2009.09.006. PMID 20402166
- [Background] Klein K, Hartman SK, Teruya J, Hui SK. An algorithmic approach to coagulation testing. Dis Mon. 2012 Aug;58(8):431-9. doi: 10.1016/j.disamonth.2012.04.006. No abstract available. PMID 22818557
- [Background] Kozek-Langenecker S, Sorensen B, Hess JR, Spahn DR. Clinical effectiveness of fresh frozen plasma compared with fibrinogen concentrate: a systematic review. Crit Care. 2011;15(5):R239. doi: 10.1186/cc10488. Epub 2011 Oct 14. PMID 21999308
- [Background] Kozek-Langenecker SA. Perioperative coagulation monitoring. Best Pract Res Clin Anaesthesiol. 2010 Mar;24(1):27-40. doi: 10.1016/j.bpa.2009.09.009. PMID 20402168
- [Background] Levi M, Schultz M, van der Poll T. Coagulation biomarkers in critically ill patients. Crit Care Clin. 2011 Apr;27(2):281-97. doi: 10.1016/j.ccc.2010.12.009. PMID 21440202
- [Background] Levi M, van der Poll T, Schultz M. Systemic versus localized coagulation activation contributing to organ failure in critically ill patients. Semin Immunopathol. 2012 Jan;34(1):167-79. doi: 10.1007/s00281-011-0283-7. Epub 2011 Jul 30. PMID 21805225
- [Background] Lisman T, Bakhtiari K, Pereboom IT, Hendriks HG, Meijers JC, Porte RJ. Normal to increased thrombin generation in patients undergoing liver transplantation despite prolonged conventional coagulation tests. J Hepatol. 2010 Mar;52(3):355-61. doi: 10.1016/j.jhep.2009.12.001. Epub 2009 Dec 24. PMID 20132999
- [Background] Lisman T, Caldwell SH, Burroughs AK, Northup PG, Senzolo M, Stravitz RT, Tripodi A, Trotter JF, Valla DC, Porte RJ; Coagulation in Liver Disease Study Group. Hemostasis and thrombosis in patients with liver disease: the ups and downs. J Hepatol. 2010 Aug;53(2):362-71. doi: 10.1016/j.jhep.2010.01.042. Epub 2010 May 12. PMID 20546962
- [Background] Meybohm P, Zacharowski K, Weber CF. Point-of-care coagulation management in intensive care medicine. Crit Care. 2013 Mar 19;17(2):218. doi: 10.1186/cc12527. No abstract available. PMID 23510484
- [Background] Northup PG, Caldwell SH. Coagulation in liver disease: a guide for the clinician. Clin Gastroenterol Hepatol. 2013 Sep;11(9):1064-74. doi: 10.1016/j.cgh.2013.02.026. Epub 2013 Mar 16. PMID 23506859
- [Background] Perner F, Petrányi Gy (szerk.): Szervátültetés. Budapest, Medicina, 2013.
- [Background] Piangatelli C, Faloia L, Cristiani C, Valentini I, Vivarelli M. Point of care perioperative coagulation management in liver transplantation and complete portal vein thrombosis. Case Rep Transplant. 2014;2014:487364. doi: 10.1155/2014/487364. Epub 2014 Feb 6. PMID 24653855
- [Background] Regan ER, Aird WC. Dynamical systems approach to endothelial heterogeneity. Circ Res. 2012 Jun 22;111(1):110-30. doi: 10.1161/CIRCRESAHA.111.261701. PMID 22723222
- [Background] Rice TW, Wheeler AP. Coagulopathy in critically ill patients: part 1: platelet disorders. Chest. 2009 Dec;136(6):1622-1630. doi: 10.1378/chest.08-2534. PMID 19995764
- [Background] Schaden E, Saner FH, Goerlinger K. Coagulation pattern in critical liver dysfunction. Curr Opin Crit Care. 2013 Apr;19(2):142-8. doi: 10.1097/MCC.0b013e32835ebb52. PMID 23400090
- [Background] Sohal AS, Gangji AS, Crowther MA, Treleaven D. Uremic bleeding: pathophysiology and clinical risk factors. Thromb Res. 2006;118(3):417-22. doi: 10.1016/j.thromres.2005.03.032. Epub 2005 Jul 1. PMID 15993929
- [Background] Solomon C, Sorensen B, Hochleitner G, Kashuk J, Ranucci M, Schochl H. Comparison of whole blood fibrin-based clot tests in thrombelastography and thromboelastometry. Anesth Analg. 2012 Apr;114(4):721-30. doi: 10.1213/ANE.0b013e31824724c8. Epub 2012 Feb 7. PMID 22314689
- [Background] Tahlan A, Ahluwalia J. Factor XIII: congenital deficiency factor XIII, acquired deficiency, factor XIII A-subunit, and factor XIII B-subunit. Arch Pathol Lab Med. 2014 Feb;138(2):278-81. doi: 10.5858/arpa.2012-0639-RS. PMID 24476525
- [Background] Thakur M, Ahmed AB. A Review of Thromboelastography. Int J Periop Ultrasound Appl Technol. 2012; 1 (1):25-29.
- [Background] Thorsen K, Ringdal KG, Strand K, Soreide E, Hagemo J, Soreide K. Clinical and cellular effects of hypothermia, acidosis and coagulopathy in major injury. Br J Surg. 2011 Jul;98(7):894-907. doi: 10.1002/bjs.7497. Epub 2011 Apr 20. PMID 21509749
- [Background] Tripodi A, Chantarangkul V, Primignani M, Fabris F, Dell'Era A, Sei C, Mannucci PM. The international normalized ratio calibrated for cirrhosis (INR(liver)) normalizes prothrombin time results for model for end-stage liver disease calculation. Hepatology. 2007 Aug;46(2):520-7. doi: 10.1002/hep.21732. PMID 17659574
- [Background] van Meurs M, Wulfert FM, Knol AJ, De Haes A, Houwertjes M, Aarts LP, Molema G. Early organ-specific endothelial activation during hemorrhagic shock and resuscitation. Shock. 2008 Feb;29(2):291-9. doi: 10.1097/SHK.0b013e318145a7c1. PMID 17704730
- [Background] Warnaar N, Lisman T, Porte RJ. The two tales of coagulation in liver transplantation. Curr Opin Organ Transplant. 2008 Jun;13(3):298-303. doi: 10.1097/MOT.0b013e3282fce79d. PMID 18685321
- [Background] Wheeler AP, Rice TW. Coagulopathy in critically ill patients: part 2-soluble clotting factors and hemostatic testing. Chest. 2010 Jan;137(1):185-94. doi: 10.1378/chest.08-2535. PMID 20051403
- See also: Diacaresolution — http://www.diacaresolution.com